CLINICAL TRIAL: NCT05865665
Title: Registry Of Best Up-titration STrategies in Acute Heart Failure (ROBUST-HF): a Registry of Post-acute Heart Failure Management
Brief Title: Registry Of Best Up-titration STrategies in Acute Heart Failure
Acronym: ROBUST-HF
Status: Not yet recruiting | Type: Observational
Sponsor: Heart Initiative (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); Hôpitaux Universitaires Saint-Louis-Lariboisière (Unknown); Momentum Research, Inc. (Industry); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CHF202201
Record Dates: First submitted 2023-04-03; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Acute Heart Failure
Keywords: Disease management; Medication therapy management; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized for acute heart failure: Patients admitted for acute heart failure for at least 72 hours who are not treated with optimal doses of oral medications for HF including renin-angiotensin system inhibitors (RASI), beta-blockers (BB), and mineralocorticoid receptor antagonists (MRA) meeting all eligibility criteria including elevated NT-proBNP.

SUMMARY:
STRONG-HF showed that rapid up-titration of renin-angiotensin inhibitor (RASI), beta-blocker, and mineralocorticoid receptor antagonist (MRA) to full optimal doses within 2 weeks post-discharge from a hospital admission for acute heart failure (AHF), using frequent safety assessments, significantly reduced the 180-day risk of HF readmission or death and significantly increased 90-day quality of life regardless of left ventricular ejection fraction (LVEF). Recent evidence also suggests that initiation of angiotensin-receptor neprilysin inhibitor (ARNI) and SGLT-2 inhibitors close to the time of discharge regardless of LVEF, and iron supplementation where indicated, improve patient prognosis.

In this prospective registry of patients not treated with optimal doses of oral HF medications being discharged from an admission for AHF, ROBUST-HF, data will be collected describing their post-discharge care including the management of their oral HF medications and frequency and content of post-discharge assessments and clinical outcomes through 6 months post discharge.

DETAILED DESCRIPTION:
The registry has three main aims:

1. Describe in a multi-national multi-site registry the post-discharge care of patients with AHF, inclusive of number of post-discharge visits and their timing, care providers conducting those visits, medications prescribed to patients, follow-up exams, inclusive of labs and NT-proBNP and finally outcomes during the first 6 months post-discharge.
2. Provide professional education and resources for physicians to accelerate the initiation and up-titration of evidence-based, guideline-directed medical therapies in appropriate patients following AHF hospitalization.
3. Provide hospitals and country leaders information on patterns of care for patients discharged from an admission for acute HF by summarizing and providing benchmark data reports.

This is a prospective, multinational, multicenter, observational registry of patients admitted to hospital more than 72 hours for AHF who were not previously treated with optimal doses of GDMT for HF. Prior to enrollment of patients in the registry, participating investigators will be trained with respect to best practices for management of GDMT. Patients at participating centers who meet all eligibility criteria will be enrolled at least 72 hours following admission to hospital for AHF, and data regarding the patient's characteristics and the initial hospitalization will be collected. Data including examinations, blood test results, and prescribed medications will be collected for each post-discharge outpatient visit through 6 months post-discharge. Detail regarding any death or re-hospitalization through 6 months will be collected. Patients will be contacted by phone at 6 months to assess vital status, the occurrence of any rehospitalizations, and prescribed HF medications. Patients will be enrolled into the registry in each site in at least two blocks. Each block within site will represent a period of 4 months during which at least 15 patients will be enrolled. After the end of the 4-month enrolment period and after the enrolled patients have been followed for 6 months, data from these patients will be summarized and presented to the site. Following discussions with the sites, a second period of 4 months during which an additional at least 15 patients will be enrolled will be undertaken. Once the last patient in this enrolment period has reached 6 months follow up, data will be again summarized and presented to the site for discussion. Professional education regarding effective implementation of most recent guideline-directed medical therapy will be carried out, both before the initiation of a site and during the study, as well as after all patients in the first enrolment period and second enrolment period have reached 6 months follow-up and the data summarized and presented to the site. Efforts would include site-level discussions, country-level meetings/teleconferences and global meetings/teleconferences. Educational efforts will be aimed at providing the most up to date cardiovascular science and guidelines and best practice sharing to facilitate the transfer of knowledge into practice; as well as highlighting performance gaps and providing strategies to improve that performance driving to improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the hospital for acute heart failure (diagnosed by dyspnea at rest and pulmonary congestion on chest X-ray or lung ultrasound) more than 72 hours prior to enrolment.
2. All measures within 24 hours prior to enrolment of systolic blood pressure ≥ 100 mmHg, and of heart rate ≥ 60 bpm.
3. The last measurement during the hospital admission prior to enrolment of serum potassium ≤ 5.0 mEq/L (mmol/L).
4. The last measuremet during the hospital admission prior to enrolment of NT-proBNP > 1,500 pg/mL
5. At admission and at the time of enrolment being prescribed: (1) none to < ½ the optimal dose (per the protocol) of renin angiotensin system inhibitor (RASi) - angiotensin converting enzyme inhibitor (ACEi), angiotensin receptor blocker (ARB), or angiotensin receptor-neprilysin inhibitor (ARNI), AND (2) none to < ½ the optimal dose of beta-blocker (BB), AND (3) none to ≤ ½ the optimal dose of mineralocorticoid receptor antagonist (MRA).
6. Written informed consent to participate in the study.

Exclusion Criteria:

1. Age < 18
2. Myocardial infarction, unstable angina or cardiac surgery, or percutaneous transluminal coronary intervention (PTCI), within 1 month prior to enrolment.
3. Presence at enrolment of any severe valvular stenosis or regurgitation in need of surgical correction.
4. Last measurement during the hospital admission prior to enrollment of eGFR < 30 mL/min/1.73m2 or history of dialysis.
5. Currently enrolled in a clinical study that mandates a schedule of follow-up visits for heart failure, or particular assessments or treatment for heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 5000 patients in up to 60 countries in Europe, the United States, Asia, Africa, and Latin America, in up to 300 sites globally. Patients admitted for acute heart failure for at least 72 hours who are not treated with optimal doses of oral medications for HF including renin-angiotensin system inhibitors (RASI), beta-blockers (BB), and mineralocorticoid receptor antagonists (MRA) who meet all the inclusion criteria and none of the exclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Characteristics of patients admitted to hospital for heart failure | Baseline
  Description of characteristics of patients enrolled including demographics, general and heart failure medical history, pre-admission and discharge HF medications, vital signs and laboratory findings
Description of the HF meds prescribed at discharge, and 2 weeks, and 1, 3 and 6 months with respect to optimal doses | Baseline, Week 2, Month 1, Month 3, Month 6
  Proportions of patients on any and on <½, ½-<full and ≥ full optimal doses of heart failure medication in each class (renin-angiotensin-system inhibitor or angiotensin receptor-neprilysin inhibitor, mineralocorticoid receptor antagonist, beta blocker, sodium-glucose co-transporter 2 inhibitor) at hospital discharge (baseline), and 2 weeks, 1 month, 3 months, and 6 months post hospital discharge
Risk of death through 6 months | Month 6
  Cumulative risk of all-cause death through 6 months post hospital discharge
Risk of cardiovascular death through 6 months | Month 6
  Cumulative risk of CV death through 6 months post hospital discharge
Risk of rehospitalization through 6 months | Month 6
  Cumulative risk of re-hospitalization through 6 months post hospital discharge
Risk of heart failure rehospitalization through 6 months | Month 6
  Cumulative risk of HF re-hospitalization through 6 months post hospital discharge
Risk of heart failure rehospitalization or cardiovascular death through 6 months | Month 6
  Cumulative risk of first HF re-hospitalization or CV death through 6 months post discharge
Proportion with follow-up visit within 1 week, 2 weeks, 1 month, 3 months, 6 months post discharge | Week 1, Week 2, Month 1, Month 3, Month 6
  Proportion of patients with 1 or more follow-up visits within 1 week, 2 weeks, and 1, 3, and 6 months post hospital discharge
Average time from discharge to first visit | Month 6
  Average number of days between discharge from the hospitalization for acute heart failure and the first outpatient visit post hospital discharge within 6 months
Average number of follow-up visits within 3 and 6 months | Month 3, Month 6
  Average number of outpatient follow-up visits within 3 and 6 months post discharge
Proportion of post-discharge visits through 6 months where laboratory values measured | Month 6
  Proportion of post-discharge visits through 6 months where laboratory values, including NT-proBNP, measured
Proportion of post-discharge visits through 6 months where vital signs measured | Month 6
  Proportion of post-discharge visits through 6 months where vital signs measured
Proportion of post-discharge visits through 6 months where clinical assessment of congestion done | Month 6
  Proportion of post-discharge visits through 6 months clinical assessments of congestion done

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, MD, Principal Investigator — Hôpitaux Universitaires Saint-Louis-Lariboisière, University Paris Diderot, Inserm 942

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data required to reach aims in an approved proposal, after de-identification, will be made available to investigators whose proposed use of the data has been approved by the study's Executive Committee. Proposals may be submitted up to 36 months after study completion and should be directed to the study's Principal Investigator
Time Frame: 36 months after study completion
Access Criteria: The proposed use must be approved by the study's Executive Committee.

REFERENCES:
- [Background] Bhatt DL, Szarek M, Steg PG, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Voors AA, Metra M, Lund LH, Komajda M, Testani JM, Wilcox CS, Ponikowski P, Lopes RD, Verma S, Lapuerta P, Pitt B; SOLOIST-WHF Trial Investigators. Sotagliflozin in Patients with Diabetes and Recent Worsening Heart Failure. N Engl J Med. 2021 Jan 14;384(2):117-128. doi: 10.1056/NEJMoa2030183. Epub 2020 Nov 16. PMID 33200892
- [Background] Cotter G, Davison B, Cohen-Solal A, Freund Y, Mebazaa A. Targeting the 'vulnerable' period - first 3-6 months after an acute heart failure admission - the light gets brighter. Eur J Heart Fail. 2023 Jan;25(1):30-34. doi: 10.1002/ejhf.2754. Epub 2022 Dec 21. No abstract available. PMID 36519644
- [Background] Davison BA, Senger S, Sama IE, Koch GG, Mebazaa A, Dickstein K, Samani NJ, Metra M, Anker SD, Cleland JG, Ng LL, Mordi IR, Zannad F, Filippatos GS, Hillege HL, Ponikowski P, van Veldhuisen DJ, Lang CC, van der Meer P, Nunez J, Bayes-Genis A, Edwards C, Voors AA, Cotter G. Is acute heart failure a distinctive disorder? An analysis from BIOSTAT-CHF. Eur J Heart Fail. 2021 Jan;23(1):43-57. doi: 10.1002/ejhf.2077. Epub 2021 Jan 22. PMID 33340221
- [Background] Hicks KA, Tcheng JE, Bozkurt B, Chaitman BR, Cutlip DE, Farb A, Fonarow GC, Jacobs JP, Jaff MR, Lichtman JH, Limacher MC, Mahaffey KW, Mehran R, Nissen SE, Smith EE, Targum SL. 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol. 2015 Jul 28;66(4):403-69. doi: 10.1016/j.jacc.2014.12.018. Epub 2014 Dec 29. No abstract available. PMID 25553722
- [Background] Jaarsma T, van der Wal MH, Lesman-Leegte I, Luttik ML, Hogenhuis J, Veeger NJ, Sanderman R, Hoes AW, van Gilst WH, Lok DJ, Dunselman PH, Tijssen JG, Hillege HL, van Veldhuisen DJ; Coordinating Study Evaluating Outcomes of Advising and Counseling in Heart Failure (COACH) Investigators. Effect of moderate or intensive disease management program on outcome in patients with heart failure: Coordinating Study Evaluating Outcomes of Advising and Counseling in Heart Failure (COACH). Arch Intern Med. 2008 Feb 11;168(3):316-24. doi: 10.1001/archinternmed.2007.83. PMID 18268174
- [Background] Laveau F, Hammoudi N, Berthelot E, Belmin J, Assayag P, Cohen A, Damy T, Duboc D, Dubourg O, Hagege A, Hanon O, Isnard R, Jondeau G, Labouree F, Logeart D, Mansencal N, Meune C, Pautas E, Wolmark Y, Komajda M. Patient journey in decompensated heart failure: An analysis in departments of cardiology and geriatrics in the Greater Paris University Hospitals. Arch Cardiovasc Dis. 2017 Jan;110(1):42-50. doi: 10.1016/j.acvd.2016.05.009. Epub 2016 Dec 21. PMID 28017276
- [Background] Logeart D, Berthelot E, Bihry N, Eschalier R, Salvat M, Garcon P, Eicher JC, Cohen A, Tartiere JM, Samadi A, Donal E, deGroote P, Mewton N, Mansencal N, Raphael P, Ghanem N, Seronde MF, Chavelas C, Rosamel Y, Beauvais F, Kevorkian JP, Diallo A, Vicaut E, Isnard R. Early and short-term intensive management after discharge for patients hospitalized with acute heart failure: a randomized study (ECAD-HF). Eur J Heart Fail. 2022 Jan;24(1):219-226. doi: 10.1002/ejhf.2357. Epub 2021 Oct 21. PMID 34628697
- [Background] Mamas MA, Sperrin M, Watson MC, Coutts A, Wilde K, Burton C, Kadam UT, Kwok CS, Clark AB, Murchie P, Buchan I, Hannaford PC, Myint PK. Do patients have worse outcomes in heart failure than in cancer? A primary care-based cohort study with 10-year follow-up in Scotland. Eur J Heart Fail. 2017 Sep;19(9):1095-1104. doi: 10.1002/ejhf.822. Epub 2017 May 3. PMID 28470962
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Background] Morrow DA, Velazquez EJ, DeVore AD, Desai AS, Duffy CI, Ambrosy AP, Gurmu Y, McCague K, Rocha R, Braunwald E. Clinical Outcomes in Patients With Acute Decompensated Heart Failure Randomly Assigned to Sacubitril/Valsartan or Enalapril in the PIONEER-HF Trial. Circulation. 2019 May 7;139(19):2285-2288. doi: 10.1161/CIRCULATIONAHA.118.039331. No abstract available. PMID 30955360
- [Background] Ponikowski P, Kirwan BA, Anker SD, McDonagh T, Dorobantu M, Drozdz J, Fabien V, Filippatos G, Gohring UM, Keren A, Khintibidze I, Kragten H, Martinez FA, Metra M, Milicic D, Nicolau JC, Ohlsson M, Parkhomenko A, Pascual-Figal DA, Ruschitzka F, Sim D, Skouri H, van der Meer P, Lewis BS, Comin-Colet J, von Haehling S, Cohen-Solal A, Danchin N, Doehner W, Dargie HJ, Motro M, Butler J, Friede T, Jensen KH, Pocock S, Jankowska EA; AFFIRM-AHF investigators. Ferric carboxymaltose for iron deficiency at discharge after acute heart failure: a multicentre, double-blind, randomised, controlled trial. Lancet. 2020 Dec 12;396(10266):1895-1904. doi: 10.1016/S0140-6736(20)32339-4. Epub 2020 Nov 13. PMID 33197395
- [Background] Public Policy Committee, International Society of Pharmacoepidemiology. Guidelines for good pharmacoepidemiology practice (GPP). Pharmacoepidemiol Drug Saf. 2016 Jan;25(1):2-10. doi: 10.1002/pds.3891. Epub 2015 Nov 5. No abstract available. PMID 26537534
- [Background] Van Spall HGC, Lee SF, Xie F, Oz UE, Perez R, Mitoff PR, Maingi M, Tjandrawidjaja MC, Heffernan M, Zia MI, Porepa L, Panju M, Thabane L, Graham ID, Haynes RB, Haughton D, Simek KD, Ko DT, Connolly SJ. Effect of Patient-Centered Transitional Care Services on Clinical Outcomes in Patients Hospitalized for Heart Failure: The PACT-HF Randomized Clinical Trial. JAMA. 2019 Feb 26;321(8):753-761. doi: 10.1001/jama.2019.0710. PMID 30806695
- [Background] Voors AA, Angermann CE, Teerlink JR, Collins SP, Kosiborod M, Biegus J, Ferreira JP, Nassif ME, Psotka MA, Tromp J, Borleffs CJW, Ma C, Comin-Colet J, Fu M, Janssens SP, Kiss RG, Mentz RJ, Sakata Y, Schirmer H, Schou M, Schulze PC, Spinarova L, Volterrani M, Wranicz JK, Zeymer U, Zieroth S, Brueckmann M, Blatchford JP, Salsali A, Ponikowski P. The SGLT2 inhibitor empagliflozin in patients hospitalized for acute heart failure: a multinational randomized trial. Nat Med. 2022 Mar;28(3):568-574. doi: 10.1038/s41591-021-01659-1. Epub 2022 Feb 28. PMID 35228754